CLINICAL TRIAL: NCT07146243
Title: Shoulder Injury Prevention in Adolescent Handball Players Based on Scandinavian Protocols: A Cluster-Randomized Controlled Trial
Brief Title: Shoulder Injury Prevention in Adolescent Handball Players Based on Scandinavian Protocols
Acronym: HBSP-HU-25
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HBSP-HU-CRCT25
Record Dates: First submitted 2025-08-13; First posted 2025-08-28 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-08

CONDITIONS: Injury Prevention; Shoulder Injuries
Keywords: overhead sport; handball; shoulder prevention; injury prevention
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Intervention Model Description: Two-armed Cluster-Randomised Controlled Trial
Masking Description: Due to the team-based cluster randomization and the nature of the intervention, masking of participants, coaches, and outcome assessors is not feasible. Entire teams are assigned to either the Swedish or the Norwegian shoulder injury prevention programme, making the intervention easily identifiable. The physiotherapists conducting the physical performance tests are aware of team allocation because they are also involved in the organization and supervision of the intervention sessions. However, the primary outcomes are objective, performance-based measures (e.g., CKCUEST, Y Balance Test-Upper Quarter, LSST, SDT, shoulder proprioception testing), which substantially reduces the potential risk of measurement bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swedish Shoulder Control Programme (Experimental): Female U18, Male U16 and Male U20 perform the physiotherapy component of the Swedish Shoulder Control Programme, excluding the throwing block, as it is designed for the off-season and the programme is implemented during the competitive season. Sessions are supervised by two physiotherapists, performed twice per week for a total of 18 weeks, before training sessions, and last approximately 15 minutes each.
  Interventions: Behavioral: Swedish Shoulder Control Programme
- Norwegian OSTRC Shoulder Injury Prevention Programme (Experimental): Female U16, Female U20 and Male U18 perform the Norwegian Shoulder Injury Prevention Programme (OSTRC). This evidence-based programme includes warm-up and strengthening exercises targeting the shoulder complex, designed to reduce the risk of shoulder injuries. Sessions are supervised by two physiotherapists, performed twice per week for a total of 18 weeks, before training sessions, and last approximately 15 minutes each.
  Interventions: Behavioral: Norwegian OSTRC Shoulder Injury Prevention Programme

INTERVENTIONS:
Behavioral: Swedish Shoulder Control Programme — An evidence-based warm-up and strengthening routine developed for handball players to reduce the risk of shoulder injuries. The physiotherapy component includes exercises for scapular control, rotator cuff strength, and shoulder mobility. The throwing block is excluded in this trial, as it is designed for the off-season and the programme is implemented during the competitive season. Exercises are performed twice per week before training sessions, last about 15 minutes, and are supervised by two physiotherapists.
  Other Names: Swedish Shoulder Control
  Arms: Swedish Shoulder Control Programme
Behavioral: Norwegian OSTRC Shoulder Injury Prevention Programme — An evidence-based warm-up and strengthening routine developed for handball players to reduce the risk of shoulder injuries. The programme focuses on exercises for scapular control, rotator cuff strength, and functional shoulder stability. Exercises are performed twice per week before training sessions, last about 15 minutes, and are supervised by two physiotherapists.
  Other Names: OSTRC Shoulder Injury Prevention Programme; Oslo Sports Trauma Research Centre Shoulder Programme
  Arms: Norwegian OSTRC Shoulder Injury Prevention Programme

SUMMARY:
This cluster-randomised controlled trial will evaluate the effects of two internationally recognised shoulder injury prevention programmes - the Swedish Shoulder Control programme and the Norwegian Oslo Sports Trauma Research Center Shoulder Injury Prevention programme - on shoulder function, scapular control, and injury incidence in Hungarian adolescent handball players (U16-U20). Six elite-level teams (3 male, 3 female) from a single handball academy will be randomised by cluster into two intervention arms for an 18-week intervention period. Primary outcomes are changes in objective shoulder function tests; secondary outcomes include self-reported function and weekly injury monitoring.

DETAILED DESCRIPTION:
This study is a two-armed cluster-randomised controlled trial designed to assess the effects of two established, evidence-based shoulder injury prevention programmes in Hungarian adolescent elite handball players. Both programmes have previously demonstrated effectiveness in reducing the incidence of shoulder injuries in overhead athletes; however, it remains unclear how they compare in their ability to improve specific objective outcomes such as shoulder stability, proprioception, strength, and scapular control. The trial will be conducted at a single elite handball academy, including six teams (three male, three female) in the U16-U20 age categories. Teams will be randomised at the cluster level (team) into one of two intervention arms, each performing one of the two prevention programmes for the entire competitive half-season (18 weeks).

Unlike most injury prevention studies in adolescent athletes, this trial combines weekly self-reported monitoring of shoulder health (OSTRC-O Shoulder Module) with a comprehensive battery of objective, instrumented assessments of shoulder function, scapular control, strength, and proprioception. This dual approach allows for a more precise evaluation of programme effectiveness, capturing both perceived and measurable physical changes.

This prevention trial forms part of a larger, ongoing research programme investigating shoulder function and return-to-sport readiness following shoulder injury in overhead athletes. The same battery of objective tests (scapular dyskinesis assessment, LSST, mLSST, CKCUEST, YBT-UQ, proprioception testing, isometric strength testing) used here is also applied in the broader project, allowing the present study to generate insights that directly inform both preventive strategies and post-injury rehabilitation protocols.

The findings from this trial are expected to inform refinements of existing shoulder injury prevention protocols, enhance compliance strategies, and support sport-specific adaptations for adolescent elite handball players and other overhead athletes.

ELIGIBILITY:
Inclusion Criteria:

* Registered competitive handball players from the participating academy team (U16, U18, U20; male and female).
* Age between 13 and 19 years at baseline assessment.
* Currently participating in regular handball training and matches (minimum 3 training sessions per week).
* Member of a team assigned to the intervention for the full study period.
* Provided written informed consent (and parental consent for participants under 18 years).

Exclusion Criteria:

* Acute shoulder injury at baseline preventing training
* Shoulder surgery in last 6 months
* Contraindication to resistance training
* Concurrent enrolment in another interventional study targeting the shoulder/upper limb.
* Refusal of informed consent (and parental consent for participants <18 years).

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 137 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Scapular Dyskinesis Test (SDT) - classification during flexion and abduction | Baseline and 18 weeks
  Description: Standard Kibler/McClure SDT with five consecutive repetitions of active shoulder flexion and abduction at a metronome cadence. Participants hold hand weights scaled to body mass: 1.5 kg if body mass <68.1 kg, and 2.5 kg if ≥68.1 kg. Testing is video-recorded. Two trained assessors, rate each shoulder from the videos as none / subtle / obvious dyskinesis for each plane. Primary outcome: proportion with any dyskinesis (subtle+obvious) by plane; secondary: shift in severity category from baseline. Lower prevalence/severity indicates improvement.
  Rater reliability plan: Inter-rater agreement will be quantified using weighted Cohen's kappa per plane.
Change in Y Balance Test - Upper Quarter (composite reach, % limb length) | Baseline and 18 weeks
  Description: YBT-UQ performed for each arm in three directions (medial, inferolateral, superolateral), three valid trials per direction. Composite reach score = (sum of the 3 maximal reaches / limb length) × 100. Limb length = C7 to tip of middle finger. Primary score is the composite % per arm; higher is better.
Shoulder proprioception error in external and internal rotation (absolute error, degrees) | Baseline and 18 weeks
  Joint position sense was assessed in supine position using a wrist-mounted digital angle gauge. For external rotation testing, the participant actively moved the arm to their individual full external rotation in 90° abduction. The target angle was then calculated using the formula:
  (Full ER in degrees-90)/2+90 This yields a mid-range position between neutral and the individual's maximal external rotation.
  First, with eyes open, then vision was occluded using a towel, and the procedure was repeated three times per limb: the assessor passively positioned the arm at the target, returned it to vertical, and the participant attempted to reposition it to the same angle without visual feedback.
  The absolute repositioning error (in degrees) between the target and reproduced positions was recorded for each trial, then averaged across the three trials per limb.
  Internal rotation target angle calculated as: 90-(90-Full IR in degrees)/2 Lower error values indicate better proprioceptive acuity
OSTRC-O Shoulder Module severity score (0-100) | Weekly for 18 Weeks
  Weekly Oslo Sports Trauma Research Center Overuse Injury Questionnaire (4 items). Composite 0-100 severity (higher = worse). Report mean weekly severity, prevalence of any problem (non-minimum response on any item), and prevalence of substantial problem (moderate/severe reduction in training/performance or complete inability to participate), as per standard methodology.

SECONDARY OUTCOMES:
Change in CKCUEST performance (touch count) | Baseline and 18 weeks
  Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST). Participants assume a standard push-up position with two parallel tape lines placed at a distance equal to 1.5 × the participant's biacromial breadth (measured between the lateral edges of the acromion processes). They alternately touch the opposite hand with one hand for three trials of 15 seconds each, with 30 seconds rest.
  Two outcomes are recorded:
  1. Touch count - mean number of valid touches across the three trials (per participant). Higher values indicate better upper-extremity closed-chain stability and power.
  2. Error count - number of form faults (e.g., loss of plank, hip rotation >45°, line misses) summed across the three trials. Lower values indicate better movement quality/control.
  A trained assessor records both outcomes according to published protocols, flagging invalid repetitions and documenting errors in real time.
Lateral Scapular Slide Test (LSST) total asymmetry score (3 positions) | Baseline and 18 weeks
  LSST performed by measuring the side-to-side difference (mm) in the distance between the inferior angle of the scapula (angulus inferior) and the nearest midline spinous process in three standardized arm positions: (1) arms relaxed at sides; (2) hands on hips with thumbs posterior; (3) 90° humeral abduction with internal rotation. The total LSST score is calculated as the sum of absolute asymmetries across the three positions. Lower scores indicate better scapular symmetry/control. Measurements are taken with a non-elastic, millimeter-scale measuring tape, with the athlete standing in a relaxed posture, feet shoulder-width apart.
Modified LSST (mLSST; 2 kg and 4 kg) | Baseline and 18 weeks
  Modified Lateral Scapular Slide Test (mLSST) performed in a static 30° scaption position while holding dumbbells of 2 kg and 4 kg, respectively. For each load, the side-to-side difference (mm) between the inferior angle of the scapula (angulus inferior) and the nearest midline spinous process is measured using a non-elastic, millimeter-scale measuring tape. The outcome for each load is the absolute asymmetry (mm). Lower values indicate better scapular symmetry/control under load.
Change in isometric shoulder strength - external and internal rotation | Baseline and 18 weeks
  Maximal isometric shoulder external rotation (ER) and internal rotation (IR) strength measured using a ForceFrame testing system (VALD Performance). Testing was performed in supine position with the shoulder in 90° abduction and neutral rotation. For each rotation direction, participants completed two maximal-effort trials per limb (due to time constraints; standard protocols recommend three), with ~30 seconds rest between trials.
  The highest peak force (N) from the two trials was used for analysis. Participants received standardized verbal encouragement during each trial. The ForceFrame system was calibrated before testing and measurements were recorded according to manufacturer guidelines.
Training/match exposure (minutes per week) | Weekly for 18 Weeks
  Self-reported weekly minutes of handball training, match play, and strength/conditioning. Used to adjust analyses and to compute injury rates (exploratory).
Programme adherence (sessions/week) | Weekly for 18 Weeks
  Number of completed prevention sessions per week (team logs + player self-report). Outcome: mean sessions/week per athlete and per team; proportion achieving ≥2 sessions/week.
Programme compliance (perceived usefulness score) | Weekly for 18 Weeks
  Weekly self-reported perception of the programme's usefulness on a 0-10 scale (0 = not useful at all, 10 = extremely useful). Report mean weekly score and trends over time. Used to explore the relationship between perceived usefulness and adherence.
Time-loss shoulder injury incidence (per 1,000 exposure hours) - exploratory | Up to 18 Weeks
  Any acute or overuse shoulder complaint causing time-loss (missed full training/match), verified with staff logs. Rate = injuries / 1,000 h (training + match).
Adverse events related to prevention sessions | Up to 18 Weeks
  Number and nature of adverse events (e.g., exacerbation of pain leading to missed session; other exercise-related events) recorded by staff.

CONTACTS AND LOCATIONS:
Overall Officials: Attila Pavlik, MD, PhD, Principal Investigator — Department of Sports Medicine
Locations (1):
- Handball Academy, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. Data sharing is not planned in order to comply with data protection regulations and to safeguard participant confidentiality.

REFERENCES:
- [Background] Asker M, Hagglund M, Walden M, Kallberg H, Skillgate E. The Effect of Shoulder and Knee Exercise Programmes on the Risk of Shoulder and Knee Injuries in Adolescent Elite Handball Players: A Three-Armed Cluster Randomised Controlled Trial. Sports Med Open. 2022 Jul 14;8(1):91. doi: 10.1186/s40798-022-00478-z. PMID 35834139
- [Background] Tooth C, Gofflot A, Schwartz C, Croisier JL, Beaudart C, Bruyere O, Forthomme B. Risk Factors of Overuse Shoulder Injuries in Overhead Athletes: A Systematic Review. Sports Health. 2020 Sep/Oct;12(5):478-487. doi: 10.1177/1941738120931764. Epub 2020 Aug 6. PMID 32758080
- [Background] Andersson SH, Bahr R, Clarsen B, Myklebust G. Preventing overuse shoulder injuries among throwing athletes: a cluster-randomised controlled trial in 660 elite handball players. Br J Sports Med. 2017 Jul;51(14):1073-1080. doi: 10.1136/bjsports-2016-096226. Epub 2016 Jun 16. PMID 27313171
- [Background] Clarsen B, Myklebust G, Bahr R. Development and validation of a new method for the registration of overuse injuries in sports injury epidemiology: the Oslo Sports Trauma Research Centre (OSTRC) overuse injury questionnaire. Br J Sports Med. 2013 May;47(8):495-502. doi: 10.1136/bjsports-2012-091524. Epub 2012 Oct 4. PMID 23038786